CLINICAL TRIAL: NCT04183088
Title: Regorafenib Plus Tislelizumab as First-line Systemic Therapy for Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Regorafenib Plus Tislelizumab as First-line Systemic Therapy for Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 201911021MIFB
Record Dates: First submitted 2019-11-25; First posted 2019-12-03 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — regorafenib; tislelizumab

STUDY DESIGN:
Intervention Model Description: This trial consists of 2 parts. Part 1 is a single-arm study. Part 2 of this trial is a randomized study. Subjects will be 1:1 randomized to 2 treatment groups: (1) regorafenib + tislelizumab combination regimen as used in Part 1, versus (2) regorafenib therapy. For subjects in the group 2, when imaging evaluation of tumor response indicates stable disease or progressive disease, according to RECIST v1.1, study treatment will be shifted to regorafenib + tislelizumab combination regimen.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking is None (open label) and the allocation is N/A for part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Tislelizumab intravenously + regorafenib orally (Experimental): Part 1 is a single-arm study. All eligible patients will receive tislelizumab 200 mg intravenously on day 1 every 3 weeks plus regorafenib orally 80 mg per day.
  Interventions: Drug: Tislelizumab+regorafenib for part 1;Tislelizumab+regorafenib for group 1 of part 2; Regorafenib for group 2 of part 2.
- Groups (1) of part 2: Tislelizumab intravenously + regorafenib (Experimental): Tislelizumab 200 mg intravenously on Day 1+Regorafenib its dosage in the randomized cohort will be determined according to results in the safety cohort.
  Interventions: Drug: Tislelizumab+regorafenib for part 1;Tislelizumab+regorafenib for group 1 of part 2; Regorafenib for group 2 of part 2.
- Groups (2) of part 2: regorafenib (Active Comparator): Daily dose of regorafenib 80mg/day is for week 1; Daily dose of regorafenib 120mg/day is for week 2; Daily dose of regorafenib 160mg/day is for week 3; Dosing-free interval is for week 4.
  * The dose of regorafenib will not be escalated if treatment-related AE > grade 1 occurs at the previous dose level.
  * For subjects in the group 2, when imaging evaluation of tumor response indicates stable disease or progressive disease, according to RECIST v1.1, study treatment will be shifted to regorafenib + tislelizumab combination regimen.
  Interventions: Drug: Tislelizumab+regorafenib for part 1;Tislelizumab+regorafenib for group 1 of part 2; Regorafenib for group 2 of part 2.

INTERVENTIONS:
Drug: Tislelizumab+regorafenib for part 1;Tislelizumab+regorafenib for group 1 of part 2; Regorafenib for group 2 of part 2. — There will be no dose reduction for tislelizumab in this study. In the part 1(safety cohort), if the subjects do not experience grade 2 or greater regorafenib-related adverse events after 2 cycles (6 weeks) of treatment, the dosage of regorafenib may be escalated. For subjects who escalate the regorafenib dosage to Level 2, if the subjects do not experience grade 2 or greater regorafenib-related adverse events after 2 cycles of study drug treatment, the dosage of regorafenib may be further escalated to Level 3.
  During study drug treatment, dose delay/ interruption of regorafenib will be done depending on the occurrence and severity of regorafenib-related adverse events. After dose reduction of regorafenib, if the subjects tolerate the reduced dose of regorafenib well, the investigators may consider re-escalation of regorafenib to the previous dose level, depending on the types and severity of adverse events that led to dose reduction.
  Other Names: Stivarga, BAY-73-4506, BGB-A317

SUMMARY:
Combination of anti-angiogenic molecular targeted therapy and anti- programmed cell death -1 immune checkpoint inhibitor (ICI) therapy has shown promising antitumor activity in multiple cancer types, including patients with advanced hepatocellular carcinoma (HCC). The safety profile and optimal dosage of targeted therapy should be carefully evaluated by clinical trials. Regorafenib is one of the standard second-line systemic therapy for advanced HCC. The present study will test the safety and efficacy of combination of regorafenib and tislelizumab, an anti-programmed cell death-1 ICI. The investigator(s) thus hypothesized that combination of tislelizumab and regorafenib is a tolerable regimen and may improve treatment efficacy for patients with advanced HCC. The present study will explore safety and efficacy of the combination of tislelizumab plus regorafenib as first-line therapy for advanced HCC.

DETAILED DESCRIPTION:
Combination of ICI with anti-angiogenic therapy has been most extensively studies in patients with renal cell carcinoma, for whom both ICI and anti-angiogenic therapy have proven anticancer activity as single-agent therapy. Objective response rate of 30-60% was observed, far exceeding the response rate of single-agent therapy (around 20%). Results from several early-phase trials of this type of combination also support the potential anti-tumor synergy between ICI and anti-angiogenic therapy (multi-kinase inhibitors or monoclonal antibody targeting the vascular endothelial growth factor signaling pathway) in advanced HCC. Further studies should focus on identifying the optimal targeted agent and its biologically effective dosage to achieve the best therapeutic window for the treatment of HCC.

Current evidence indicated the following:

1. Combination of ICI and anti-angiogenic therapy in advanced HCC may have better anti-tumor efficacy compared with single-agent therapy;
2. The immune modulatory effects of the multi-kinase inhibitors may be achieved at dosage lower than recommended for single-agent therapy in the clinic; using this lower dosage when combined with ICI may lower the treatment-related adverse events.
3. Objective response of 40% to 50% was recently reported in a phase 1 study of regorafenib plus nivolumab for patients with advanced gastric or colorectal cancer was reported recently (Fukuoka S, et al. American Society Of Clinical Oncology 2019, abstract#2522). Grade 3 or greater treatment-related adverse events were found in 27% of subjects who received regorafenib 80 mg per day and in 44% of patients who received regorafenib 120 mg per day. Therefore, regorafenib 80 mg/day was defined as the optimal dosage in combination with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Age ≥ 20 years, according to local regulation in Taiwan, at time of signing Informed Consent Form.
3. Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology.
4. Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies
5. Agreement to have a new tumor biopsy for eligibility to this study
6. No prior systemic therapy (including systemic investigational agents) for HCC.
7. For patients with chronic hepatitis B virus (HBV) infection: agreement to receive anti-HBV treatment (per local standard of care; e.g., entecavir) prior to study entry and willingness to continue treatment for the length of the study.
8. At least one measurable (per RECIST 1.1) lesion. Patients who received prior local therapy (e.g., radiofrequency ablation or transarterial chemoembolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1.
9. The liver tumors, if any, should occupy ≤ 50% of estimated liver volume.
10. Eastern Cooperative Oncology Group Performance Status of 0 or 1 within 7 days prior to first dose of study drug treatment.
11. Child-Pugh class A within 14 days prior to first dose of study drug treatment.
12. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to first dose of study drug treatment, unless otherwise specified:

    * Absolute neutrophil count≥1.5 * 109/L without granulocyte colony-stimulating factor support; platelet count ≥75 *109/L without transfusion; and hemoglobin≥(9 g/dL (patients may be transfused to meet this criterion).
    * Liver transaminases (AST and ALT) ≤5 x upper limit of normal (ULN)
    * Serum creatinine ≤1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
    * Urine dipstick for proteinuria < 2+ (within 7 days prior to initiation of study treatment). Patients who have ≥ 2+ proteinuria on dipstick urinalysis at baseline will be eligible if he/she have daily protein excretion of < 1 g documented by a 24-hour urine collection.
13. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, ≥ 8 weeks after the last dose of regorafenib, and ≥ 120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test ≤ 7 days of first dose of study drug treatment.
14. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study, ≥ 8 weeks after the last dose of regorafenib, and ≥ 120 days after the last dose of tislelizumab

Exclusion Criteria:

1. Histological diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
2. Liver tumor(s) with main portal vein thrombosis.
3. Known human immunodeficiency virus (HIV) infection.
4. History of esophageal/gastric varices or active peptic ulcers that are considered to have high risk of bleeding.
5. History of upper gastrointestinal bleeding within 1 year.
6. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs."
7. Prior allogeneic stem cell or solid organ transplantation.
8. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
9. Prior therapy with an anti-Programmed cell death protein(PD)-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte protein 4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
10. Local therapy to liver (e.g., radiofrequency ablation, transarterial chemoembolization, etc.) within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure.
11. Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to initiation of study treatment, except for palliative radiotherapy to bone lesions. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
12. Patients with a history of treated and, at the time of screening, asymptomatic central nervous system(CNS) metastases are eligible, provided they meet all the following:

    * Brain imaging at screening shows no evidence of interim progression
    * Have measurable disease outside the CNS
    * No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
    * No stereotactic radiation or whole-brain radiation within 14 days prior to randomization,
    * Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases.
    * Following treatment, these patients may then be eligible, provided all other criteria, including those for patients with a history of brain metastases, are met.
13. Active autoimmune diseases or history of autoimmune diseases that may relapse. Patients with the following diseases are not excluded and may proceed to further screening: vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
14. History of drug-induced pneumonitis or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
15. Known active tuberculosis or other active infection.
16. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment. Core biopsy or other minor surgical procedure within 3 days prior to the first dose of regorafenib.
17. History of malignancy other than HCC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival(OS) rate> 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer.
18. Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen) may be allowed.
19. Current or recent (within 10 days of first dose of study treatment) use of aspirin (>325 mg/day), other anti-platelet therapy (e.g., dipyramidole, ticlopidine, clopidogrel, and cilostazol), or full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose.
20. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment.
21. Uncontrolled hypertension: systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg despite anti-hypertension medications ≤ 28 days before randomization or first dose of drug
22. Any of the following cardiovascular risk factors:

    * Conditions occurring ≤ 28 days before first dose of study drug treatment: Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, symptomatic pulmonary embolism, any episode of syncope or seizure.
    * Conditions occurring ≤ 6 months before first dose of study drug treatment: any history of acute myocardial infarction, any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV, any event of ventricular arrhythmia ≥ Grade 2 in severity, any history of cerebrovascular accident
23. Concurrent participation in another therapeutic clinical study.
24. Was administered a live vaccine ≤ 4 weeks before first dose of study drug treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety cohort: 14 participants with treatment related serious adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) V5.0. | Day 1, Change from Day 1 to 23-37 days after the last dose of study drug treatment.
  14 or fewer participants who experience grade 3 or greater treatment-related adverse events at the 80 mg per day level, as defined by Common Terminology Criteria for Adverse Events (CTCAE)V5.0.
Randomized cohorts: Objective response rate (ORR) (co-primary) | about 1 year
  The percentage of 100 participants with radiologically complete or partial response as determined by the investigator according to Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Randomized cohorts: Progression-free survival (PFS) (co-primary) | about 1 year
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Safety cohort: safety as assessed by 25 participants experiencing who incidence and severity of total AE, liver related AE, and immune-related AE. | Day 1, Change from Day 1 to 23-37 days after the last dose of study drug treatment.
  25 participants experiencing who incidence and severity of total AE, liver related AE, and immune-related AE.as defined by Common Terminology Criteria for Adverse Events (CTCAE)V5.0.
Safety cohort: Proportion of 25 participants who may escalate the dose of regorafenib (continuous dosing) during study drug treatment | Day 1 of each cycle
  An adequate supply of regorafenib will be dispensed to participants on Day 1 of each new cycle (once every 3 weeks). Each time study drug is dispensed, compliance will be evaluated and encouraged. Treatment compliance will also be monitored by drug accountability log.
Safety cohort: Objective response rate (ORR) | about 1 year
  The percentage of 25 participants with radiologically complete or partial response as determined by the investigator according to both RECIST 1.1 and the immune-RECIST.
Randomized cohort: safety as assessed by 100 participants experiencing who incidence and severity of total AE, liver related AE, and immune-related AE. | Day 1, Change from Day 1 to 23-37 days after the last dose of study drug treatment.
  100 participants experiencing who incidence and severity of total AE, liver related AE, and immune-related AE.as defined by Common Terminology Criteria for Adverse Events (CTCAE)V5.0.
Randomized cohort: Objective response rate (ORR) | about 1 year
  The percentage of 100 participants with radiologically complete or partial response as determined by the investigator according to both RECIST 1.1 and the immune-RECIST.
Safety cohort: progression-free survival (PFS) | about 1 year
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 and the immune-RECIST or death from any cause (whichever occurs first).
Randomized cohort: progression-free survival (PFS) | about 1 year
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 and the immune-RECIST or death from any cause (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan